CLINICAL TRIAL: NCT03991442
Title: A Randomized, Double-blind, Multicenter, Phase III Study to Evaluate the Efficacy and Safety of BR1010 in Essential Hypertension Patients Who do Not Adequately Respond to Fimasartan/Amlodipine Combination
Brief Title: BR1010 in Patients With Essential Hypertension Patients Who do Not Adequately Respond to Fimasartan/Amlodipine Combination
Acronym: FINAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR-FAHC-CT-301
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR1010 and Fimasartan/Amlodipine placebo (Experimental): BR1010 or Fimasartan/Amlodipine
  Interventions: Drug: Fimasartan/Amlodipine
- BR1010 placebo and Fimasartan/Amlodipine (Active Comparator): BR1010 or Fimasartan/Amlodipine
  Interventions: Drug: Fimasartan/Amlodipine

INTERVENTIONS:
Drug: Fimasartan/Amlodipine — Active Comparator: a fixed dose combination of Fimasartan/Amlodipine or placebo
  Other Names: BR1010 or placebo

SUMMARY:
The objective of this clinical study is to evaluate the efficacy and safety by comparing the BR1010 treatment group to the fimasartan/amlodipine treatment group at Week 8 in patients with essential hypertension who do not adequately respond to Fimasartan/Amlodipine combination

ELIGIBILITY:
Inclusion Criteria:

1.Voluntarily provided a written consent to participate in this clinical study 2.19 years old or above Koreans living in Korea 3.Patients with uncontrolled essential hypertension at screening time(Visit 1)

* Use antihypertensive drugs:140 mmHg ≤ sitSBP < 200 mmHg
* Naïve: 160 mmHg ≤ sitSBP < 200 mmHg 4.Patients with uncontrolled hypertension after Fimasartan/Amlodipine 30/5mg treatment for 4 weeks at randomization(Visit 2) (Selected Arm:140 mmHg ≤ sitSBP < 200 mmHg 5.Able to understand this study, be cooperative in the execution of the study, and participate in the study until its completion

Exclusion Criteria:

1. Difference of SiSBP ≥ 20 mmHg and SiDBP ≥ 10 mmHg in 3 blood pressure measurements in the selected reference arm at the screening visit
2. Blood pressure results showing sitDBP ≥ 120 mmHg at screening and baseline visit(Visit 1; Both Arm, Visit 2: Selected Arm)
3. Treatment Compliance of Fimasartan/Amlodipine 30/5mg < 70%
4. Heart failure(New York Heart Association class 3 and 4), ischemic heart disease, peripheral vascular disease
5. Percutaneous Coronary Artery within 6 months prior to study
6. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter; or other arrhythmia conditions that are determined to be clinically significant by the investigator
7. Patients who have history of severe cerebrovascular disease within 6 months prior to study
8. Type I Diabetes Mellitus or Uncontrolled Type II Diabetes Mellitus(HbA1c > 9% at screening visit
9. Patients who have history of severe or malignant retinopathy within 6 months prior to study
10. Pregnant or lactating women
11. Planning pregnancy during the study period or have childbearing potential but are not using acceptable contraceptive methods
12. Patients taking other clinical trial drugs within 4 weeks from the time of visit for screening
13. Patients who are judged unsuitable to participate in this study by investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
sitting systolic blood pressure | 8weeks from Baseline Visit
  The change of sitting systolic blood pressure

SECONDARY OUTCOMES:
sitting systolic blood pressure | 2weeks and 4weeks from Baseline Visit
  The change of sitting systolic blood pressure
sitting systolic blood pressure and sitting diastolic blood pressure | 2weeks, 4weeks and 8weeks from Baseline Visit
  The change of sitting systolic blood pressure and sitting diastolic blood pressure
The ratio of subjects who get normalized blood pressure | 2weeks, 4weeks and 8weeks from Baseline Visit
  The ratio of subjects who get normalized blood pressure
Response Rate | 2weeks, 4weeks and 8weeks from Baseline Visit
  Response Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Boryung Pharmaceutical Co., Ltd, Seoul, South Korea